CLINICAL TRIAL: NCT00376701
Title: Combination Therapy in Neovascular Age-Related Macular Degeneration (AMD): A Three-armed, Randomized, Prospective Clinical Trial of Low Fluence Photodynamic Therapy(rPDT) With Adjunctive Avastin and Triamcinolone Acetonide (Kenalog)(Triple Therapy) Versus rPDT With Adjunctive Avastin (Double Therapy) Versus Monotherapy With Avastin.
Brief Title: Combination Therapy for Age-Related Macular Degeneration.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: QLT Inc. (Industry); Canadian Retinal Trials Group (Other)
Responsible Party: Principal Investigator, Thomas G. Sheidow, Vitreoretinal Surgeon, Associate professor of Ophthalmology, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R-06-441; Health Canada Control #106990; 9427-U0207/2-21C
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Age Related Macular Degeneration
Keywords: Choroidal Neovascularization; Photodynamic Therapy; Age Related Macular Degeneration; Triamcinolone Acetonide; Avastin; Visudyne
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Reduced fluence PDT plus intravitreal Kenalog (2 mg) plus intravitreal Avastin 1.25 mg
  Interventions: Drug: Avastin (Bevacizumab); Drug: Bevacizumab
- 2 (Experimental): Reduced fluence PDT plus intravitreal Avastin
  Interventions: Drug: Avastin (Bevacizumab); Drug: Bevacizumab
- 3 (Experimental): Intravitreal Avastin and sham reduced fluence PDT
  Interventions: Drug: Avastin (Bevacizumab); Drug: Bevacizumab

INTERVENTIONS:
Drug: Avastin (Bevacizumab) — Avastin 1.25 mg intravitreal
Drug: Bevacizumab — Intravitreal 1.25 mg
  Other Names: Avastin
  Arms: 1
Drug: Bevacizumab — Intravitreal 1.25 mg
  Other Names: Avastin
  Arms: 2
Drug: Bevacizumab — Intravitreal Avastin 1.25 mg and sham reduced fluence PDT
  Other Names: Avastin
  Arms: 3

SUMMARY:
The primary purpose of the study is to investigate whether patients with Choroidal Neovascularization secondary to Age-related Macular Degeneration, receiving triple or double therapy compared to monotherapy with Avastin will reduce the intervention rate with equivalent safety and efficacy.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the leading cause of irreversible blindness in developed countries throughout the world.The beneficial therapeutic effect of Photodynamic Therapy (PDT)in the treatment of AMD is modest. The treatment benefit of PDT may be moderated by PDT-induced, non-selective effects in the choroidal circulation (resulting in hypoxia-induced stimulation of angiogenesis through increased vascular endothelial growth factor (VEGF)production), direct injury to the retinal pigment epithelium, and subretinal fluid/hemorrhage or post-treatment inflammation secondary to PDT. There is potential that supplemental Avastin (through VEGF inhibition) or intravitreal Triamcinolone Acetonide (ITA) treatments (through non-specific membrane stabilizing, anti-neovascular, and anti-inflammatory activities) could minimize the effect of these processes, enhancing the efficacy of PDT. Presently, PDT, the current gold standard,in combination with Avastin and/or Kenalog is being more widely used in exactly this fashion and may become the standard of care without the necessary randomized clinical trial. However, the treatment benefit of these interventions is uncertain as is their safety profile.

This randomized, controlled trial addresses the potential supplemental therapeutic effect of intravitreal injection of Triamcinolone Acetonide and/or Avastin in conjunction with photodynamic therapy for the treatment of sub-foveal CNVM secondary to AMD.

ELIGIBILITY:
Inclusion Criteria:

1. Choroidal neovascularization (CNV) secondary to age-related macular. All lesion subtypes, based upon IVFA evaluation will be included.
2. CNV under the geometric centre of the foveal avascular zone.
3. Evidence of choroidal neovascular activity as suggested by one of the following: sub-retinal lipid, sub-retinal hemorrhage, and documented loss of 3 lines of vision within the last three months.
4. Greatest linear dimension of the lesion </= 5400 um.
5. Visual acuity of between 20/32 and 20/800 in the study eye - Equivalent to Early Treatment of Diabetic Retinopathy Study (ETDRS) eye chart score of 5 to 75 letters at 2 metres.
6. Willingness and ability to participate and provide written informed consent

Exclusion Criteria:

1. Individuals with choroidal neovascularization from causes other than AMD.
2. Individuals physically unable to tolerate intravenous fluorescein angiography or Verteporfin injections. (Specifically, individuals with inadequate venous access or an allergy/sensitivity to fluorescein dye/porphyrins will be excluded.)
3. Any intraocular surgery within 3 months in the study eye.
4. Prior retinal or vitreous surgery including posterior segment vitrectomy or scleral buckling in the study eye.
5. Any significant ocular disease that has compromised or could compromise vision in the study eye and confound analysis of the primary outcome.
6. Individuals with physical or mental disabilities that prevent accurate vision testing.
7. History of treatment of CNV in study eye other than extrafoveal confluent laser photocoagulation.
8. Prior photodynamic therapy for CNV in the study eye.
9. Active hepatitis or clinically significant liver disease
10. Any patient with recent history of new onset cardiac disease or thromboembolic CNS event in the past.
11. Subjects who are in an experimental therapy study or who have received experimental therapy within the last 12 weeks.
12. Subjects who are a poor medical risk because of other systemic diseases or active uncontrolled infections.
13. Women of child-bearing potential who are not on two forms of effective contraception during the trial and for at least 60 days following the last dose of study medications.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2006-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To investigate whether patients with CNV secondary to AMD, receiving triple or double therapy compared to monotherapy with Avastin, will reduce the intervention rate with equivalent safety and efficacy. | 1 year

SECONDARY OUTCOMES:
To compare between treatment groups: | 1 year
Whether combination therapy with rPDT + iA and rPDT + iAK in patients with sub-foveal CNVM of all types secondary to ARMD will result in a significant improvement in visual acuity defined as 2 or more lines (10+ letters) on a standardized ETDRS chart c | 1 year
Lesion growth and activity over the study period. | 1 year
Contrast sensitivity. | 1 year
The rate of cataract progression. | 1 year
Central retinal thickness via Optical Coherence Tomography (OCT). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G. Sheidow, MD, Principal Investigator — The University of Western Ontario
Locations (5):
- Canada (5):
  - The University of Alberta and Capital Health, Edmonton, Alberta
  - The University of British Columbia, Vancouver, British Columbia
  - Dr. Stanley G. Shortt, Victoria, British Columbia
  - Ivey Eye Institute, St. Joseph's Health Care Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario